CLINICAL TRIAL: NCT01217268
Title: Use of Telemedicine in Collaboration Between a Psychogeriatric Unit and Nursing
Brief Title: Use of Telemedicine in Collaboration Between a Psychogeriatric Unit and Nursing Homes
Acronym: TESAM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Morten Lang-Ree, CEO, Sykehuset Innlandet Health Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TESAM
Record Dates: First submitted 2010-09-22; First posted 2010-10-08 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2011-05

CONDITIONS: Dementia; Behavioural Disorders
MeSH Terms: conditions — Dementia; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Training and supervision of staff (Experimental): Staff members get training in person centered care by supervision using video-conference kit
  Interventions: Behavioral: Training in person centered care by supervision using video-conference

INTERVENTIONS:
Behavioral: Training in person centered care by supervision using video-conference — The investigators will use video-conference for supervising and training of staff members in nursing homes

SUMMARY:
The investigators want to evaluate the use of video-conference in the collaboration between the investigators psychogeriatric department and nursing homes. The study aim is to give supervision on a regular basis to the caregivers on a special care unit for patients with dementia with behavioural disturbances during a period of half a year. The investigators want to investigate the impact on caregivers and patients by applying certain tests at baseline, during the intervention and half a year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being resident in a special care unit for persons with dementia

Exclusion Criteria:

* Shorter stay than four weeks before inclusion
* terminally ill

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric inventory - nursing home version (NPI-NH) | week 48
  The investigators want to find out if a supervision of staff members over a six months time, using video-conference technic, contributes to improvement in patients' behaviour registered by NPI-NH

SECONDARY OUTCOMES:
Person-centered Care Assessment Tool (P-CAT) Person centered care assessment tool (P-CAT) | week 48
  Measures the effect of our intervention related to apply person centred dementia care

CONTACTS AND LOCATIONS:
Overall Officials: Oskar H Sommer, PhD, Principal Investigator — SykehusetInnlandet, Norway
Locations (1):
- Sykehuset Innlandet HF, Reinsvoll, Norway